CLINICAL TRIAL: NCT07016412
Title: A Phase IIb, Randomized, Double-blind, Placebo- Controlled, Parallel Group Study to Assess the Efficacy and Safety of Ensifentrine-glycopyrrolate Fixed-dose Combination at Two Dose Levels Compared to Glycopyrrolate or Ensifentrine Monotherapy in Subjects With COPD
Brief Title: A Phase IIb Ensifentrine-glycopyrrolate Fixed-dose Combination Dose Ranging Study in Subjects With COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPL554-CO-212
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; bronchodilator; ensifentrine-glycopyrrolate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment Arm A: Ensifentrine plus Glycopyrrolate (Experimental): Ensifentrine 3 mg / Glycopyrrolate 42.5 mcg
  Interventions: Drug: Ensifentrine 3 mg; Drug: Glycopyrrolate 42.5 mcg
- Treatment Arm B: Ensifentrine plus Glycopyrrolate (Experimental): Ensifentrine 3 mg / Glycopyrrolate 21.25 mcg
  Interventions: Drug: Ensifentrine 3 mg; Drug: Glycopyrrolate 21.25 mcg
- Treatment Arm C: Glycopyrrolate (Active Comparator): Glycopyrrolate monotherapy 42.5 mcg
  Interventions: Drug: Glycopyrrolate 42.5 mcg
- Treatment Arm D: Glycopyrrolate (Active Comparator): Glycopyrrolate monotherapy 21.25 mcg
  Interventions: Drug: Glycopyrrolate 21.25 mcg
- Treatment Arm E: Ensifentrine (Active Comparator): Ensifentrine monotherapy 3 mg
  Interventions: Drug: Ensifentrine 3 mg
- Treatment Arm F: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ensifentrine 3 mg — Administered by a standard jet nebulizer, twice daily for 28 consecutive days
  Arms: Treatment Arm A: Ensifentrine plus Glycopyrrolate; Treatment Arm B: Ensifentrine plus Glycopyrrolate; Treatment Arm E: Ensifentrine
Drug: Glycopyrrolate 21.25 mcg — Administered by a standard jet nebulizer, twice daily for 28 consecutive days
  Arms: Treatment Arm B: Ensifentrine plus Glycopyrrolate; Treatment Arm D: Glycopyrrolate
Drug: Glycopyrrolate 42.5 mcg — Administered by a standard jet nebulizer, twice daily for 28 consecutive days
  Arms: Treatment Arm A: Ensifentrine plus Glycopyrrolate; Treatment Arm C: Glycopyrrolate
Drug: Placebo — Administered by a standard jet nebulizer, twice daily for 28 consecutive days
  Arms: Treatment Arm F: Placebo

SUMMARY:
This study will assess the safety and efficacy of fixed dose combinations of ensifentrine with two different glycopyrrolate dose levels compared to placebo and to the individual components of the fixed dose combinations, each administered twice a day via standard jet nebulizer, in adult subjects with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Enrolled participants will be expected to participate for approximately 7 weeks: 1 to 2 weeks for screening, 4 weeks of treatment, and 1 week of follow up. Participants will be randomized to one of 6 treatment arms: two fixed dose combinations of ensifentrine (3 mg) and glycopyrrolate (either 21.25 or 42.5 mcg), the 3 individual components as monotherapies, or placebo. All treatments will be administered twice a day via oral inhalation by a standard jet nebulizer. The primary objective of this study is to evaluate the bronchodilator effects of the fixed dose combinations compared to each of the individual components and to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males are eligible to participate if they agree to use contraception or abstinence, and refrain from donating fresh unwashed semen during the study and for at least 30 days post-study
* Females are eligible to participate if they are not pregnant, breastfeeding and if one of the following conditions apply:

  1. Not a woman of child-bearing potential OR
  2. Agrees to follow the contraceptive guidance from screening throughout the study and for at least 30 days post-study
  3. Agrees not to donate eggs for the purpose of reproduction from screening throughout the study and for at least 30 days post-study
* Current of former cigarette smokers with a history of smoking ≥ 10 pack years at the time of signing informed consent [number of pack years = (number of cigarettes per day / 20) × number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Pipe and/or cigar use cannot be used to calculate pack-year history. Former smokers are defined as those who have stopped smoking for at least 6 months prior to signing informed consent. Smoking cessation programs are permitted during the study
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines with symptoms compatible with COPD
* A score of ≥ 2 on the Modified Medical Research Council (mMRC) Dyspnea Scale at the Screening Visit
* Post-bronchodilator (4 puffs of albuterol) spirometry during the Screening Period demonstrating both the following:

  1. FEV1/forced vital capacity (FVC) ratio of < 0.70 AND
  2. FEV1 ≥ 30 % and ≤ 70% of predicted normal
* A posterior-anterior chest x-ray (CXR) during the Screening Period or within 12 months of signing the Informed Consent Form (ICF) showing no clinically significant abnormalities unrelated to COPD. If a CXR within the past 12 months is not available but a computed tomography (CT) scan within the same time period is available, the CT scan may be reviewed in place of a CXR
* Subjects on no maintenance/background therapy or subjects on stable maintenance as either long-acting β2-agonist (LABA) or long-acting β2-agonist/Inhaled corticosteroid (LABA/ICS) therapy are eligible. Subjects taking maintenance therapy must demonstrate regular use of maintenance therapy, in any form, for at least 60 days prior to signing informed consent and agree to continue use of their current permitted LABA or LABA/ICS medication for the duration of the screening and treatment period
* Capable of withholding from short-acting bronchodilators for 4 hours prior to spirometry testing. Subjects receiving maintenance therapy with a LABA or LABA/ICS must be capable of withholding twice-daily maintenance therapy for 24 hours and once-daily maintenance therapy for 48 hours prior to initiation of any spirometry
* Capable of using the study jet nebulizer correctly
* Ability to perform acceptable spirometry in accordance with ATS/ERS guidelines
* Willing and able to attend all study visits and adhere to all study assessments and procedures

Exclusion Criteria:

* Concomitant clinically significant pulmonary disease other than COPD (i.e., asthma, tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, sleep apnea (unless controlled with stable continuous positive airway pressure [CPAP] use), known alpha-1 antitrypsin deficiency, core pulmonale or other non-specific pulmonary disease
* Within 6 months prior to randomization, a COPD exacerbation requiring hospitalization
* Within 3 months prior to randomization, use of oral or systemic therapies for COPD exacerbations (for example, oral, intravenous, or intramuscular glucocorticoids, antibiotics, theophylline, and roflumilast)
* History of life-threatening COPD, including Intensive Care Unit admission and/or requiring intubation
* Severe comorbidities including

  1. unstable cardiac disease (myocardial infarction within 1 year prior to randomization, unstable angina within 6 months prior to randomization, unstable or life-threatening arrhythmia requiring intervention within 3 months prior to randomization, diagnosis of New York Heart Association (NYHA) class III or IV heart disease, or
  2. any other clinically significant medical conditions including uncontrolled diseases (e.g., endocrine, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric [e.g. untreated significant depression, anxiety or history of suicidality], or ophthalmic diseases) that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject
* History of or clinically significant on-going bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within 6 months prior to randomization
* History of narrow angle glaucoma
* History of hypersensitivity or intolerance to aerosol medications, albuterol, ensifentrine, or glycopyrrolate or any of its excipients/components, anticholinergic agents, or sympathomimetic amines
* History of or current malignancy of any organ system, treated or untreated within the 5 years prior to randomization, except for localized basal or squamous cell carcinoma of the skin
* Other significant psychiatric disease that would likely result in the subject not being able to complete the study, in the opinion of the Investigator
* Findings on physical examination that an investigator considers to be clinically significant or abnormal during the Screening Period including hematology, biochemistry, viral serology, and ECG
* Prior or current use of Ohtuvayre (ensifentrine)
* Previous lung resection or lung reduction surgery within 1-year of randomization
* Long term oxygen use defined as oxygen therapy prescribed for greater than 12 hours per day. As needed oxygen use (≤ 12 hours per day) is not exclusionary
* Pulmonary rehabilitation unless such treatment has been stable from 4 weeks prior to signing the ICF and plans to remain stable during the study. Pulmonary rehabilitation programs should not be started or completed during participation in the study
* Major surgery (requiring general anesthesia) in the 6 weeks prior randomization, lack of full recovery from surgery at randomization, or planned surgery through the end of the study
* Current or history of drug or alcohol abuse within the 5 years prior to randomization
* Estimated glomerular filtration rate (eGFR) < 30 mL/min as tested during the Screening Period
* Alanine aminotransferase (ALT) ≥ 2 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≥ 2 × ULN, alkaline phosphatase and/or total bilirubin > 1.5 × ULN (subjects with Gilbert's syndrome can be included with total bilirubin >1.5 × ULN as long as direct bilirubin is ≤ 1.5 × ULN)
* Use of an experimental drug within 30 days or 5 half-lives of signing the ICF, whichever is longer, and/or participation in a study treatment-free follow-up phase of a clinical study within 30 days prior to signing the ICF
* Use of an experimental medical device or participation in a follow-up phase of an experimental medical device clinical study within 30 days prior to informed consent
* Affiliation with the investigator site, including an Investigator, Sub-Investigator, study coordinator, study nurse, other employee of participating investigator or study site or a family member of the aforementioned

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in average forced expiry volume in 1 second (FEV1) area under the curve versus time, from time 0 to 4 hours (AUC0-4h) | Baseline and Days 1, 14, 28, and 29

SECONDARY OUTCOMES:
Change from baseline in peak FEV1 measured over 4 hours post-dose | Baseline and Day 28
Change from baseline in average FEV1 area under the curve versus time, from time 0 to 12 hours (AUC0-12h) | Baseline and Day 28
Change from baseline in morning trough FEV1 on Day 29 | Baseline and Day 29
Change from baseline in evening trough FEV1 on Day 28 | Baseline and Day 28
Change from baseline in morning trough FEV1 on Day 28 | Baseline and Day 28
Change from baseline in average FEV1 AUC0-4h measured after first dose on Day 14 | Baseline and Day 14
Change from baseline in peak FEV1 measured over 4 hours after first dose on Day 14 | Baseline and Day 14
Change from baseline in average FEV1 AUC0-4h measured after first dose on Day 1 | Baseline and Day 1
Change from baseline in peak FEV1 measured over 4 hours after first dose on Day 1 | Baseline and Day 1
Change in symptoms of dyspnea as measured by Transition Dyspnea Index (TDI) | Days 14 and 28
Change from baseline in health-related quality of life as measured by Saint George's Respiratory Questionnaire (SGRQ) total score | Baseline and Day 28
Incidence of treatment emergent adverse events (TEAEs) | From first dose through end of study (approximately 5 weeks)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - SEC Clinical Research, LLC, Dothan, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Downtown LA Research Center Inc - ClinEdge, Los Angeles, California
  - California Medical Research Associates, Inc., Northridge, California
  - Northern California Research Corp, Sacramento, California
  - Clinical Research of West Florida Inc, Clearwater, Florida
  - Fleming Island Center For Clinical Research, Fleming Island, Florida
  - Florida Institute For Clinical Research LLC, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of West Florida Inc - Tampa, Tampa, Florida
  - Centricity Research Columbus Georgia, Columbus, Georgia
  - Southeast Lung Associates Research, Rincon, Georgia
  - ASHA Clinical Research - Hammond, Hammond, Indiana
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research, Rockville, Maryland
  - Revive Research Institute, Inc, Southfield, Michigan
  - Midwest Clinical Research LLC, St Louis, Missouri
  - The Clinical Research Center LLC - CRN, St Louis, Missouri
  - Sierra Clinical Research, Las Vegas, Nevada
  - Trialfinity Clinical Research Center, Hamilton, New Jersey
  - Horizon Family Medical Group, New Windsor, New York
  - American Health Research Inc, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Stern Research Partners, LLC, Huntersville, North Carolina
  - Monroe Biomedical Research -343 Venus St, Monroe, North Carolina
  - Carolina Research Center, Inc, Shelby, North Carolina
  - Remington Davis Clinical Research, Columbus, Ohio
  - Advance Clinical Research, Dayton, Ohio
  - Velocity Clinical Research - Anderson - PPDS, Anderson, South Carolina
  - Pharmacorp Clinical Trials Incorporated, Charleston, South Carolina
  - Piedmont Research Partners LLC, Fort Mill, South Carolina
  - Velocity Clinical Research - Gaffney - PPDS, Gaffney, South Carolina
  - Lowcountry Lung and Critical Care PA, North Charleston, South Carolina
  - Monroe Biomedical Research Charleston, North Charleston, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Velocity Clinical Research - Union, Union, South Carolina
  - Chattanooga Research & Medicine, Chattanooga, Tennessee
  - ClinSearch - Chattanooga, Chattanooga, Tennessee
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - MultiSpecialty Clinical Research, Inc, Johnson City, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - Corsicana Medical Research, Corsicana, Texas
  - Houston Pulmonary Sleep & Allergy Associates, Cypress, Texas
  - Greater Heights Memorial Pulmonary and Sleep, Houston, Texas
  - Houston Pulmonary Medicine Associates, PA, Houston, Texas
  - Huntsville Research Institute LLC, Huntsville, Texas
  - Element Research Group, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Tranquil Clinical Research, Webster, Texas

IPD SHARING:
Plan to Share IPD: No